CLINICAL TRIAL: NCT06276426
Title: Plants Optimizing Development Study
Brief Title: Plants Optimizing Development Study (PODS)
Acronym: PODS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Soy Nutrition Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24468
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Healthy Children
Keywords: soy; isoflavones; cognition; body composition; fecal microbiota; metabolic risk
MeSH Terms: interventions — Soy Foods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy (Experimental): The experimental group will be asked to consume 2 servings/day of soy foods for 3 months
  Interventions: Other: Soy foods
- Non-Soy Plant-Based Foods (Active Comparator): The control group will be asked to consume 2 servings/day of non-soy plant-based foods for 3 months
  Interventions: Other: Non-Soy Plant-Based Foods

INTERVENTIONS:
Other: Soy foods — Soy milk, soy yogurt, tofu, tempeh, soy nuts, edamame, soy protein bar, and soy-based frozen meat substitutes.
  Arms: Soy
Other: Non-Soy Plant-Based Foods — Pea milk, almond milk yogurt, chickpeas, chickpea chips, lentil chips, non-soy protein bar, and non-soy based frozen meat substitutes.
  Arms: Non-Soy Plant-Based Foods

SUMMARY:
This study aims to conduct a randomized clinical trial to measure the effects of a 3-month daily mixed-soy food intervention vs. a control group receiving isocaloric foods on reproductive hormones, body composition, metabolic risk, fecal microbiota, and cognition among 8-11-year-old children. Additionally, this study will assess soy food intake immediately following participation in the clinical trial to determine changes in soy food acceptance in children.

DETAILED DESCRIPTION:
The central hypothesis is that greater soy isoflavone consumption does not alter sex steroid levels but is associated with beneficial clinical outcomes of body composition, metabolic health, and gut-brain axis among pre- and early adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Child assent and parent/guardian consent
* Free of any food allergy
* 8-11 years of age
* Tanner scale score of ≤ 2
* 20/20 or corrected vision
* No antibiotic usage in the past 3 months
* ≤1 serving/d of soy food habitual consumption

Exclusion Criteria:

* Non-assent or consent by child assent and/or parent/guardian
* Presence of any food allergy
* Younger than 8 years or older than 11 years
* Presence of specific neurological and genetic disorders (i.e., Autism, Cerebral Palsy, Multiple Sclerosis, Down syndrome)
* Presence of endocrine, metabolic, and gastrointestinal disease e.g., hypertension, diabetes, celiac disease
* Tanner scale score of > 2
* Not 20/20 or uncorrected vision
* Antibiotic usage in the past 3 months
* >1 serving/d of soy food habitual consumption

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Sex steroid excretion | 3 months (Baseline vs Follow-up)
  urinary concentration of androgen and estrogenic steroids

SECONDARY OUTCOMES:
Gut microbiota | 3 months (Baseline vs Follow-up)
  Gut microbiota will be assessed using a fecal sample. Outcomes will include α-diversity/community richness and evenness (Shannon Index), β-diversity (microbial structures), and Firmicutes:Bacteroidetes ratio.
Attentional Accuracy | 3 months (Baseline vs Follow-up)
  Changes in accuracy (%) between groups using a computerized flanker task.
Attentional Reaction Time | 3 months (Baseline vs Follow-up
  Changes in reaction time (ms) between groups using a computerized flanker task.
Hippocampal-dependent Relational memory | 3 months (Baseline vs Follow-up)
  Spatial memory task accuracy.
Body Composition | 3 months (Baseline vs Follow-up)
  DXA scans will be used to assess whole body bone density and Android:Gynoid ratio.
Metabolic Markers | 3 months (Baseline vs Follow-up)
  Fasted venous blood will be collected from the antecubital vein of the arm to measure TG, LDL, HDL, TC, and FG using the Piccolo Xpress Analyzer (Abaxis, Inc.).
Pubertal Staging | 3 months (Baseline vs Follow-up)
  Tanner pubertal stage will be assessed using the Growing and Changing Questionnaire. The survey consists of line drawings23 representing the Tanner stages for genital size and for pubic hair and to record which drawing most closely represents the child's stage.
Cognitive Abilities and Academic Achievement | 3 months (Baseline vs Follow-up)
  Woodcock Johnson Tests of Cognitive Abilities and Academic Achievement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided